CLINICAL TRIAL: NCT01541241
Title: Uterine Haemodynamic Changes in Patients With Copper Intrauterine Device Induced Bleeding
Brief Title: Study About Patients Using Copper Intrauterine Device
Acronym: IUD
Status: Completed | Type: Observational
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Other Study IDs: Ayman-1
Record Dates: First submitted 2012-02-14; First posted 2012-02-29 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Copper Intrauterine Device Induced Bleeding
Keywords: Intrauterine contraceptive device (IUD) is one of the most frequently used methods of birth control around the world; Uterine Hemodynamic changes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- copper IUD used: Group I: includes 50 cases using CIUD and complaining of menorrhagia or menometrorrhagia.
  Group II: includes 50 cases using CIUD and not complaining of abnormal uterine bleeding.

SUMMARY:
THE AIM OF THE this study is to assess the hemodynamic changes of uterine artery in patients with CIUD induced bleeding by using transvaginal color Doppler indices (uterine artery resistance index and pulsatility index) to prove the relationship between these changes and bleeding in these patient .

DETAILED DESCRIPTION:
Intrauterine contraceptive device (IUD) is one of the most frequently used methods of birth control around the world. IUD induced irregular uterine bleeding is one of the main problems for many women using this method. In the first year of insertion of the IUDs, between 5 to 15% of women will have their IUDs removed because of bleeding. The use of IUD has been unfortunately associated with functional failure on one hand, and medical complications on the other hand. Despite the increasing use of intrauterine device, their further dissemination has been limited by high expulsion rates and the withdrawal of their use for medical reasons, mainly bleeding and pain.

Following insertion of modern copper IUD, menstrual blood loss increases by about 55%, and this level of bleeding continues for the duration of IUD use. These changes occur more rapidly, and iron supplementation is recommended.

There are several possible mechanisms that explain the cause of excessive bleeding in patients using IUD. Several studies reported that IUD insertion increase the production of prostaglandins in the endometrium which cause increased vascularity, vascular permeability, and inhibit platelet activity and therefore increase menstrual bleeding.

Recent studies have reported that IUD causes cyclo-oxygenase-2 (COX-2) up expression, the subsequent elevated prostanoid biosynthesis and signaling can promote the expression of pro-angiogenic factors, such as vascular endothelial growth factor (VEGF) , basic fibroblast growth factor (bFGF), platelet derived growth factor (PDGF), angioprotein-1 (Ang-1) and angioprotein-2 (Ang-2) or down-regulate the expression of anti-angiogenic genes such as cathepsin-D.

There are several mechanisms explaining the association of the pulsatility index (PI) and resistance index (RI) of uterine artery with menstrual blood loss. It has been suggested that menorrhagia, may be caused by an increased uterine secretion of prostanoids leading to impaired haemostasis.

Temporary post-insertion rise in prostaglandin concentrations coincided with the phase of increased bleeding and pain. There is over expression of mRNA and protein of COX-2 enzyme leading to overproduction of prostaglandins in the endometrium after the insertion of copper intrauterine device (CIUD).

Other vasoactive substances may also be involved, including nitric oxide (NO) which is a potent vasodilator produced the vascular endothelium. NO is present in the human endometrium and myometrium.

There is evidence that NO may play a part in acute and chronic inflammation. The introduction of intrauterine device into the uterine cavity induces a foreign body reaction in the surrounding endometrium. NO is present in the foreign body inflammatory reaction around loosened joint replacement implants. Thus, it is possible that IUD also induces NO synthesis in the surrounding tissue. There is also a connection between NO synthesis and prostaglandin synthesis. NO directly interacts with COX, which is responsible for prostaglandin synthesis and causes an increase in enzymatic activity.

There are also other possible mechanisms explaining the association of the PI of uterine artery with menstrual blood loss. Women with menorrhagia show a significant increase in endothelial cell proliferation, reflecting disturbed angiogenesis.

It is possible that there are also other vascular abnormalities resulting from disturbed angiogenesis. In abnormal vessels, poor contractibility and dysfunction of the haemostatic system may cause menorrhagia and decreased impedance. The expression of VEGF and its receptor, kinase insert domain-containing receptor (KDR) and microvessel density (MVD) were increased in endometrium after using CIUD.

Based on these findings, uterine artery Doppler indices RI, PI were widely investigated in order to identify the uterine hemodynamic changes in patients with IUD induced bleeding.

The protocol for this study will be approved by the local ethics committee, and informed consent will be obtained from the patients.

Every woman will be subjected to the following:

* Complete history taking including age, parity, duration of CIUD use, timing of insertion of CIUD, history of other contraception method before insertion of CIUD, menstrual history before and after CIUD insertion including duration and amount of menstrual flow, regularity and length of the cycle, history of any drug intake, blood disease and any medical disorders were considered.
* Clinical examination including general, abdominal, and pelvic examination.
* Ultrasound examination will be done .After instructing the patients to empty their bladders, transvaginal ultrasound will done with the woman in the supine position with her legs semi-flexed and abducted to allow for easy manipulation of the vaginal probe at different angles with the application of the push-pull technique. A coupling gel will applied to the vaginal probe which was then introduced into a rubber glove and another layer of coupling gel was applied to the glove. The probe will then introduced into the vagina for systematic scanning.

Ultrasound examination will done on cycle days 2-5 unless there was continual bleeding, using a 7.5 MHz transvaginal transducer with color Doppler facilities . All the ultrasound measurements were measured between 9:00 and 11:00 am to eliminate diurnal variation.

The uterus and the ovaries will first visualized using conventional B-mode ultrasound to check the uterine size, the dimensions of its walls, presence of uterine masses and the accurate placement of the device inside the uterus.

Blood flow indices of the uterine artery will then calculated to obtain the pulsatility index (PI) and the resistance index (RI) according to the following equations: PI = (A - B)/mean, and RI = (A - B)/A, where A is the peak systolic, B is the end-diastolic Doppler shift, and the mean is the maximum Doppler shift frequency taken over the cardiac cycle. The mean PI and RI will calculated by combining three waveforms of the left and right uterine artery and were used for subsequent statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Regularly menstruating women before CIUD insertion.
2. Age between 18 and 35 years.
3. Hormonal treatment has not been taken at least two months before the study.
4. Non steroidal anti-inflammatory drugs has not been taken 24 hours before the examination.

Exclusion Criteria:

1. Pregnancy.
2. The presence of pelvic pathology as ovarian cysts, pelvic endometriosis, endometrial polyps or fibrosis.
3. Present or past history of pelvic inflammatory disease.
4. Patients on hormonal treatment in the last two months before the study.
5. Patients on non steroidal anti-inflammatory drugs last 24 hours before the examination.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic, hospital out patient clinic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2012-02-28 (Actual); Study Completion 2012-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Abdelazim Elgamal, Residant, Principal Investigator — Shoubra General Hospital
Locations (1):
- Shoubra Maternity Hospital, Cairo, Shoubra, Egypt